CLINICAL TRIAL: NCT04398485
Title: A Phase 1 Study of ION251 Administered by Intravenous Infusion to Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of ION251 Administered to Patients With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ION251-CS1
Record Dates: First submitted 2020-05-11; First posted 2020-05-21 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
Keywords: multiple myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ION251 (Experimental): In Part 1, the dose escalation phase, increased amounts of ION251 will be administered at multiple time points by intravenous (IV) infusion during 28-day cycles. In Part 2, the determined RP2D of ION251 will be administered at multiple time points by IV infusion.
  Interventions: Drug: ION251

INTERVENTIONS:
Drug: ION251 — ION251 administered by IV infusion

SUMMARY:
The purpose of this study is to determine the maximum-tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of ION251 in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a two-part, multi-center first in human study of ION251 in up to 80 participants. Part 1 will use a 3+3 dose-escalation scheme in sequential cohorts to determine the MTD and RP2D during repeated 28-day treatment cycles. MTD will be determined by the number of participants with AEs meeting the dose-limiting toxicity (DLT) criteria during Cycle 1. The MTD determined in Part 1 will be used with other variables to inform a RP2D for participants proceeding to Part 2 for further assessments in the safety, tolerability and anti-myeloma activity.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at the time of informed consent
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Measurable multiple myeloma (MM)
4. In need of systemic treatment for MM and either is refractory to or has failed treatment with, is intolerant to or has refused, or is not otherwise a candidate in the opinion of the Investigator, for any of the currently available established therapies known to provide clinical benefit in relapsed/refractory MM. Refractory to treatment is defined as documented MM disease progression while on or within 60 days from the last dose (LD) of treatment

Exclusion Criteria:

1. Screen laboratory results as follows, or any other clinically significant abnormalities in screen laboratory values that would render a participant unsuitable for inclusion

   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN)
   * Total bilirubin > 1.3 × ULN
   * Absolute neutrophil count ≤ 1.0 1000/cubic millimeter (k/mm^3)
   * Platelet count < 50 k/mm^3
   * Hemoglobin < 8.0 g/dL
   * Estimated glomerular filtration rate (eGFR) < 50 milliliters per minute (mL/min)/1.73 square meter (m^2)
   * Urine albumin creatinine ratio > 100 mg/g
2. History of or current plasma cell leukemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, and skin changes) syndrome, solitary bone or extramedullary plasmacytoma as the only evidence for plasma cell dyscrasia, myelodysplastic syndrome or a myeloproliferative neoplasm
3. Uncontrolled hypertension (systolic pressure ≥ 160 mm of mercury (mm Hg) and/or diastolic pressure ≥ 100 mm Hg)
4. Presence of a bleeding disorder or an underlying disease state associated with active bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum-Tolerated Dose (MTD) | Up to 28 days from the last dose of study drug in Cycle 1 (each cycle is 28 days)
  MTD is defined as the maximum dose at which ≤ 1 of 3 evaluable participants experiences a dose-limiting toxicity (DLT) within Cycle 1 and there are 2 of 3 or 2 of 6 evaluable participants in the next higher-dose level experiencing a DLT within Cycle 1. If no dose in the dose-escalation has 2 of 3 or 2 of 6 evaluable participants experiencing a DLT, the highest dose level is considered the MTD
Recommended Phase 2 Dose (PR2D) | Up to 28 days from the last dose of study drug
  RP2D is chosen based on the dose response and exposure-response analyses of the pooled clinical PK, PD, safety results, and anti-myeloma activity from both Part 1 and Part 2

SECONDARY OUTCOMES:
Safety and Tolerability as Measured by the Incidence of TEAEs | Up to 28 days from the last dose of study drug
Incidence of Abnormal Laboratory Values and Vital Signs | Up to 28 days from the last dose of study drug
Cmax: Maximum Observed Concentration ION251 | From Baseline up to 28 days from the last dose of study drug
AUC[0-t]: Area Under the Plasma Concentration-Time Curve from Hour zero to t of ION251 | From Baseline up to 28 days from the last dose of study drug
t1/2: Distribution Half-life of ION251 | From Baseline up to 28 days from the last dose of study drug
Trough Concentration of ION251 | From Baseline up to 28 days from the last dose of study drug
Urine 0-24 Hour (hr) Excretion of ION251 | Up to 12 months from the last dose of study drug

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Rrmc, Los Angeles, California
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mondala PK, Vora AA, Zhou T, Lazzari E, Ladel L, Luo X, Kim Y, Costello C, MacLeod AR, Jamieson CHM, Crews LA. Selective antisense oligonucleotide inhibition of human IRF4 prevents malignant myeloma regeneration via cell cycle disruption. Cell Stem Cell. 2021 Apr 1;28(4):623-636.e9. doi: 10.1016/j.stem.2020.12.017. Epub 2021 Jan 20. PMID 33476575